CLINICAL TRIAL: NCT06384157
Title: A Phase II Double Blind, Placebo Controlled, Randomised, Dose-Ranging Study to Assess the Safety and Efficacy of INDV-2000 Over 3 Months in Treatment Seeking Individuals With Opioid Use Disorder
Brief Title: Proof of Concept and Dose-ranging Study of INDV-2000 in Individuals With Moderate to Severe Opioid Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INDV-2000-201
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, double-blind, placebo-controlled study where the investigator, assessor, sponsor and participant are masked.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 100 mg INDV-2000 QD dosed by two 50 mg extended-release tablets (Experimental)
  Interventions: Drug: INDV-2000
- 200 mg INDV-2000 QD dosed by two 100 mg extended-release tablets (Experimental)
  Interventions: Drug: INDV-2000
- 400 mg INDV-2000 QD dosed by two 200 mg extended-release tablets (Experimental)
  Interventions: Drug: INDV-2000
- Placebo dose (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: INDV-2000 — INDV-2000 is a highly potent and selective OX1R antagonist that is being developed as a therapy for the treatment of OUD.
  Arms: 100 mg INDV-2000 QD dosed by two 50 mg extended-release tablets; 200 mg INDV-2000 QD dosed by two 100 mg extended-release tablets; 400 mg INDV-2000 QD dosed by two 200 mg extended-release tablets
Other: Placebo — This is a randomized, double-blind, placebo-controlled study.
  Arms: Placebo dose

SUMMARY:
The purpose of this study is to measure safety and efficacy and to determine dose-response relationship for INDV-2000 in participants with moderate to severe Opioid Use Disorder (OUD) who are new to treatment, have recently initiated or completed short-term medically supervised withdrawal with transmucosal (TM) buprenorphine, and are interested in transitioning to a non opioid treatment.

DETAILED DESCRIPTION:
From Day 1 to Day 7, TM buprenorphine and randomized INDV-2000/Placebo will be administered, INDV-2000/Placebo will be administered alone from Day 8 onward. The randomized treatment period starts when the participant receives randomized treatment (at Day 1) and ends at his/her last study visit, if on INDV-2000/Placebo alone, or ends when starting buprenorphine rescue therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Participant must be 18 or the legal age of consent in the jurisdiction in which the study is taking place to 65 years of age inclusive, at the time of signing the informed consent.
  2. Able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures, be able to comply with protocol requirements, rules and regulations of study site, and be likely to complete all the study interventions.
  3. Males or females with moderate or severe opioid use disorder (OUD) by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria who are looking to transition from daily short-term opioid agonist treatment (medically supervised withdrawal) to non-opioid treatment.
  4. Have not been on medication for opioid use for 3 months prior to the current treatment episode, and satisfies either a or b below.

     1. The participant will initiate, or is undergoing medically supervised withdrawal, and

        * In the opinion of the investigator, the participant is able to achieve a stable dose of transmucosal (TM) buprenorphine between ≤24 mg inclusive prior to randomization.
        * Current opioid agonist treatment does not exceed 35 days from the start of TM buprenorphine to the end of Screening window.
     2. The participant recently completed medically supervised withdrawal outside of the study, and

        * Time elapsed between last dose of TM buprenorphine or other withdrawal medication and Study Day 1/randomization does not exceed 21 calendar days.
        * Recently completed opioid agonist treatment does not exceed 35 days of TM buprenorphine dosing days inclusive of medically assisted withdrawal dosing.
  5. Male participants who are sexually active with individuals who are of childbearing potential must agree to use a medically acceptable forms of contraception from Screening until at least 90 days after the last dose of study medication. The following methods of contraception are considered to be medically acceptable: established use of oral, injected or implanted hormonal contraception; placement of an intrauterine device or intrauterine system; or use of a double barrier method of contraception (condom or occlusive cap with use of a spermicide), or abstinence.
  6. A female participant of non-childbearing potential, or a male of childbearing potential if

     * She agrees to use a medically acceptable form of contraception from Screening until at least 90 days after the last dose of study medication. The following methods of contraception are considered to be medically acceptable: abstinence; established use or oral, injected or implanted hormonal contraception; placement of an intrauterine device or intrauterine system; or use of a double barrier method of contraception (condom or occlusive cap with use of a spermicide).
     * She is not pregnant as confirmed by a negative serum screening and or urine human chorionic gonadotrophin test on Study Day 1.
     * She is not lactating.
  7. Body mass index (BMI) within 18.0 to 40.0 kg/m2 (inclusive)

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:

  1. Have a current diagnosis, other than OUD, requiring chronic opioid treatment.
  2. Have a concurrent primary substance use disorder, as defined by DSM-5 criteria, other than opioid, tobacco, cannabis or alcohol use disorders.
  3. Meet DSM-5 criteria for severe substance use disorder other than opioids.
  4. Have a medical history of clinically significant neurological, cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, or psychiatric disorder that would impact participation in the study as judged by an Investigator or medically responsible physician.
  5. Had an opioid overdose event within the 6 months prior to the Screening Visit.
  6. Uses any substance of abuse via the injection route more than 2 times per week over the last 3 months prior to Screening.
  7. Have clinically significant abnormal biochemistry, hematology or urinalysis results that would impact participation in the study as judged by an Investigator or medically responsible physician.
  8. Have a history of narcolepsy, cataplexy, obstructive or central sleep apnea.
  9. Have disorders that may interfere with drug absorption, distribution, metabolism and excretion processes.
  10. History of suicidal ideation within 30 days prior to providing written informed consent as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale (C-SSRS) completed at the Screening Visit or history of a suicide attempt (per the C-SSRS) in the 6 months prior to informed consent.
  11. Serious cardiac illness or other cardiac assessments including, but not limited to:

      * Uncontrolled arrhythmias.
      * History of congestive heart failure.
      * Myocardial infarction <6 months from receipt of first dose of investigational medicinal product (IMP)
      * Uncontrolled symptomatic angina
      * QT interval corrected with Fridericia's formula (QTcF) >450 msec for males and >470 msec for females or history of prolonged QT syndrome.
  12. Have any combination of the following at screening:

      * Total bilirubin ≥1.5×upper limit of normal (ULN) (with direct bilirubin >1.3 mg/dL),
      * Alanine aminotransferase (ALT) ≥3×ULN
      * Aspartate aminotransferase (AST) ≥3×ULN
      * International normalized ratio (INR) >1.2 for participants not receiving anticoagulation therapy, >3.0 for participants on conventional coagulation therapy, >3.5 for participants on intensive anticoagulation, or
      * Estimated glomerular filtration rate <60 mL/min by Cockroft-Gault formula.
  13. Current symptomatic hepatic or biliary disease, including participants with cholecystectomy <90 days prior to Screening.
  14. Use of a long-acting buprenorphine or naltrexone treatment for OUD within 2 years or 1 year of the screening visit, respectively.
  15. Concurrent treatment or treatment with an investigational drug, or participation in any other clinical study within 30 days prior to the signing the informed consent form.
  16. Blood or platelets donation of greater than 500 mL within 56 days or plasma donation within 7 days of screening; clinically significant anemia or low hemoglobin (<11 g/dL for females, <12 g/dL for males).
  17. Known allergy or hypersensitivity to IMP or its excipients.
  18. Any condition that, in the opinion of an Investigator or medically responsible physician, would interfere with evaluation of the IMP or interpretation of participant safety or study results.
  19. Is a member of site staff, has a financial interest in Indivior, or is an immediate family member of anyone directly involved in the study (ie, site staff, Indivior, or Clinical Research Organization [CRO] employee).
  20. Participants who are unable, in the opinion of an Investigator or medically responsible physician, to comply fully with the study requirements, including prohibited concomitant therapies.
  21. Current incarceration, treatment for OUD required by court order, or pending incarceration/legal action that could prevent participation or compliance in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Proportion (probability) of participants without treatment failure by the end of Week 12 (Day 85). | 12 weeks
  The treatment failure is defined as meeting either one of the two criteria.
  1. Urine Drug Screen (UDS, dipstick) positive for opioids, or fentanyl on 4 consecutive assessments while participants on the Investigational Medicinal Product (IMP) (INDV-2000 or placebo) alone (after Day 8 visit).
  2. Discontinued the IMP (INDV-2000 or placebo) prematurely.

SECONDARY OUTCOMES:
Proportion (probability) of visits with opioid abstinence while participants are on IMP alone. | From Week 1 to Week 13
  Abstinence is based on negative UDS and self-report use.
Participant's percentage of visits with opioid abstinence during the whole study follow-up. | 13 Weeks
  Abstinence is based on negative UDS and self-report use.
Incidence, severity and relatedness of adverse events, treatment-emergent adverse events, serious adverse events and events leading to discontinuation and deaths. | 17 weeks
  Number of participants reporting adverse events
Opioid Craving Assessment | 13 Weeks
  7-item self-reported instrument to assess the participant's craving in the past week, on a likert scale of 1 to 7 (Strongly Disagree as 1, Disagree, Slightly Disagree, Neither Agree nor Disagree, Slightly Agree, Agree, or Strongly Agree as 7). The 7 questions assess general craving, and the following 6 dimensions: preoccupation or obsessive thoughts, anticipation of negative reinforcement, anticipation of positive reinforcement, motivation, drive and intention to use opioids, feeling lack of control or automaticity, and feeling uneasiness related to opioid use.
Cmax on Day 1 and Day 15/16 | 2 Weeks
  PK sampling are done under the PK Substudy
Tmax on Day 1 and Day 15/16 | 2 Weeks
  PK sampling are done under the PK Substudy
AUC0-24 on Day 1 and Day 15/16 | 2 Weeks
  PK sampling are done under the PK Substudy
Cavg on Day 1 and Day 15/16 | 2 Weeks
  PK sampling are done under the PK Substudy
Cmin on Day 1 and Day 15/16 | 2 Weeks
  PK sampling are done under the PK Substudy
CL/F on Day 1 and Day 15/16 | 2 Weeks
  PK sampling are done under the PK Substudy
Clinical Opiate Withdrawal Scale (COWS) score | 4 weeks
  The COWS is an 11-item, validated instrument used to assess symptoms of opiate withdrawal. The score is the sum of the response to each of the 11 items and ranges from 0 to 48. A score of 5 to 12 is considered mild, 13 to 24 is moderate, 25 to 36 is moderately severe, and a score >36 is considered severe withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Global Director Clinical Development, Study Director — Indivior Inc.
Locations (35):
- United States (35):
  - Boyett Health Services Inc, Hamilton, Alabama
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - North County Clinical Research, Oceanside, California
  - Empire Clinical Research, Pomona, California
  - Artemis Institute For Clinical Research - San Diego, San Diego, California
  - Imagine Research of Palm Beach County, Boynton Beach, Florida
  - Bold City Clinical Research, Jacksonville, Florida
  - Vitalix Kissimmee, Kissimmee, Florida
  - Accel Research Sites - Lakeland, Lakeland, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - Segal Trials Miami Lakes, Miami Lakes, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - Maryland Treatment Centers, Baltimore, Maryland
  - Vitalix Clinical, Worcester, Massachusetts
  - Insight Research Institute, Flint, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - IMA Clinical Research, Las Vegas, Nevada
  - Oasis Clinical Research, Las Vegas, Nevada
  - Richmond Behavioral Associates, Staten Island, New York
  - Dr Vando Medical Services, The Bronx, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Pahl Pharmaceutical Professionals, LLC, Oklahoma City, Oklahoma
  - SP Research PLLC Rivus Wellness and Research Insitute, Oklahoma City, Oklahoma
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Prisma Health Addiction Medicine Center, Greenville, South Carolina
  - Insite Clinical Research, LLC, DeSoto, Texas
  - El Paso Clinical Trials, El Paso, Texas
  - HD Research, Houston, Texas
  - Progressive Clinical Research Llc, Bountiful, Utah
  - Alpine Research Organisation, Clinton, Utah
  - Boeson Clinical Research, Provo, Utah